CLINICAL TRIAL: NCT05033652
Title: Impact on Mortality of Screening for Kidney Disease Associated With a Specialized Intervention During Hospitalization in a Territorial Hospital Trust
Acronym: WARNING KD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PREPS/2019/OM-01
Record Dates: First submitted 2021-07-27; First posted 2021-09-05 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Acute Kidney Injury; Chronic Kidney Diseases
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Cluster step wedge
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard strategy (No Intervention)
- Warning KD strategy (Experimental)
  Interventions: Other: WARNING KD

INTERVENTIONS:
Other: WARNING KD — Within 48h of detecting an abnormal creatinemia value (GFR<30 or AKIN2 and AKIN3), the biology laboratory will communicate the patient's information to the "WARNING KD" team. This team consists of one nephrologist and one clinical pharmacist who will trigger the initial management in the department and then, if the patient has a persistant warning signal during hospitalization, define the patient's course of treatment for discharge. Patients requiring special care will be oriented towards a nephrologist and the patient's GP will be alerted to the benefit of addressing the patient to a nephrologist for multidisciplinary management with a therapeutic project according to the recommendations for good therapeutic practices.
  Arms: Warning KD strategy

SUMMARY:
Kidney disease in its chronic or acute form shares many risk factors for initiation, progression and prognosis with an increase in morbidity and mortality, the length of hospitalization and the cost associated with stages of increasing severity. Its overall estimated prevalence in the general population is 13% and 0.5% from stage 4, for which referral to a nephrologist is recommended to reduce mortality, slow progression of renal disease and better prepare for treatment by renal replacement. Acute kidney injury (AKI) is defined as a sudden increase in serum creatinine (Scr) with a prognostic classification of increasing severity. The population with chronic kidney disease (CKD) is often hospitalized and is frequently complicated by AKI, however CKD is asymptomatic for a long time, requiring structure screening in populations at risk.

Performing Scr assays during hospitalization is an opportunity to screen patients with severe CRD or ARI requiring specialized treatment during and after hospitalization. A nephrological opinion is recommended for patients with severe CKD and AKI.

Based on preliminary studies "MRC GARD" (NCT02938611) and "ARI TARGET" (NCT03192189), the study investigators identified the frequency of patients with increased Scr corresponding to stages ≥4 of CKD and to stage1b of ARI during their hospitalization. They found that 50% of patients hospitalized with a severe AKI had a CKD prior to their hospitalization.

The use of dosages of Scr during hospitalization has been studied for AKI but without targeting high-risk subgroups and with discordant results. The study investigators plan to carry out a pragmatic study to show that an intervention combining alerts with Scr dosage to detect severe forms of CRD and AKI during hospitalization associated with the systematic intervention of a specialized dedicated team associating nephrologist and pharmacist to the scale of a GHT will improve patient and renal survival 1 year after screening.

ELIGIBILITY:
Inclusion Criteria:

* The patient or their representative must have given their free and informed consent oral consent
* The patient must be a member or beneficiary of a health insurance plan
* Patient living in the Gard, France
* Patient with abnormal dose:

  * Severe grade 4 or 5 CKD suspected in front of a GFR <30 mL / min / 1.73m2 persisting during hospitalization.
  * Acute kidney injury > stage 1 defined by an increase in serum creatinine of at least 100% in less than 7 days or a threshold greater than 354 µmol / l.

Exclusion Criteria:

* The subject is participating in another category I interventional study, or is in a period of exclusion determined by a previous study
* It is impossible to give the subject or their representative informed information
* The patient is under safeguard of justice or state guardianship
* Patient is pregnant, parturient or breastfeeding.
* Patient unable to express consent
* Patient with Stage 1 Acute kidney injury defined by an increase in serum creatinine of more than 26 µmol / l in less than 48 hours or a 50% increase in serum creatinine within 7 days.
* Patient with stage 1 to 3 CKD (glomerular filtration rate (GFR)> 30 mL / min / 1.73m2)

  * Palliative/end-of-life patients
  * Patients who died within 72 hours of receiving the signal
  * Patients hospitalized in nephrology after an emergency room visit only
  * Patients under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1680 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-12-16 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Mortality | 12 Months
  Information taken from national database

SECONDARY OUTCOMES:
Need for renal support | 12 Months
  yes / no. Information available in the SNDS database and the REIN register.
Mortality | 30 days
  Information taken from national database
Emergency start of renal support management | 12 Months
  Yes/no with exact date noted if yes. Information available in the REIN register
Oriented of patient towards autonomous support techniques | 12 Months
  Yes/no. Information available in the REIN register
Which autonomous support techniques used | 12 Months
  renal transplant or home dialysis
Use of an arteriovenous fistula during the first session | 12 Months
  Yes/no
Duration of initial hospitalization | 12 Months
  Days
Duration of rehospitalizations | 12 Months
  Days
Causes of rehospitalizations | 12 Months
  Information taken from SNDS database
The rate of patients with stage ≥4 CKD followed by a nephrologist | 12 Months
  Data-collection via the medical file on visit(s) to the nephrologist during hospitalization; after discharge from hospital via data collected in the SNDS database
Rate of patients with at least one inappropriate drug prescription for renal function | Inclusion
Rate of patients with at least one inappropriate drug prescription for renal function | 3 Months
Rate of patients with at least one inappropriate drug prescription for renal function | 12 Months
Prevalence of drug prescriptions slowing down the progression of the kidney disease and treating complications | Inclusion
Prevalence of drug prescriptions slowing down the progression of the kidney disease and treating complications | 3 Months
Prevalence of drug prescriptions slowing down the progression of the kidney disease and treating complications | 12 Months
Estimation of the incremental cost-efficiency ratio | 12 Months
  ratio of la difference in cost and the difference in life expectancy between the two strategies
National scale estimation of costs avoided | 12 Months
  Total costs of healthcare consumption and the cost of setting up the device in the two management strategies
Evaluation of the satisfaction carers of patients in the interventional group during hospitalization | end of the interventional strategy phase (minimum 3 months, maximum 12 months)
  6-item custom questionnaire on 5-point Likert scale with free comment section
Evaluation of the satisfaction doctors of patients in the interventional group during hospitalization | end of the interventional strategy phase (minimum 3 months, maximum 12 months)
  5-item custom questionnaire on 5-point Likert scale with free comment section
Evaluation of the satisfaction doctors of patients in the interventional group during hospitalization | 12 Months
  5-item custom questionnaire on 5-point Likert scale with free comment section
Evaluation of patient satisfaction of patients in the interventional group | end of the interventional strategy phase (minimum 3 months, maximum 12 months)
  3-item custom questionnaire on 5-point Likert scale free comment section
Evaluation of patient satisfaction of patients in the interventional group | 12 months
  3-item custom questionnaire on 5-point Likert scale free comment section
Evaluate the implementation of the "WARNING KD" management model at individual facilities according to the Template for Intervention Description and Replication (TIDieR) checklist. | Over the study - maximum 2 years
  12-item checklist

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Moranne, Principal Investigator — CHU Nimes
Locations (3):
- France (3):
  - CH Alès Cévennes, Alès
  - CH Bagnols-sur-Cèze, Bagnols-sur-Cèze
  - CHU de Nîmes, Nîmes